CLINICAL TRIAL: NCT03473821
Title: Motor Imagery to Facilitate Sensorimotor Relearning (MOTIFS) After ACL Injury: A Randomized Controlled Trial
Brief Title: Motor Imagery to Facilitate Sensorimotor Relearning After ACL Injury
Acronym: MOTIFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2016/413
Record Dates: First submitted 2018-02-28; First posted 2018-03-22 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL Injury; Return to Sport; Mental Training; Dynamic Motor Imagery; Anterior Cruciate Ligament; Knee Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Intervention Model Description: 1:1 single assessor-blinded adaptive randomized controlled trial, which will conform to the CONSORT statement
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded, but due to the nature of the study, neither the primary investigator, participant, nor the care providers can be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training (No Intervention): Participants in this group will undergo rehabilitation for ACL injury consisting of neuromuscular training according to care-as-usual treatment common to physical therapy professionals.
- MOTIFS (Experimental): Participants in this group will receive an intervention that has been developed according to our new training model, known as MOTor Imagery to Facilitate Sensorimotor re-learning (MOTIFS). In this intervention, patients will receive a neuromuscular training rehabilitation program with integrated dynamic motor imagery.
  Interventions: Behavioral: MOTIFS

INTERVENTIONS:
Behavioral: MOTIFS — o MOTor Imagery to Facilitate Sensorimotor re-learning (MOTIFS) is an individualized and physical activity-specific integrated model that includes aspects of both neuromuscular training, as used in rehabilitation practices, and Dynamic Motor Imagery (DMI). DMI is a form of mental training in which the participant images him-/herself performing a task from a first-person perspective in order to maximize functional equivalence to the task in question. This includes dynamic, physical movement, as well as mental imaging. The intervention provides a framework for designing individualized, physical activity-specific rehabilitation exercises for knee-injured people.
  Other Names: Neuromuscular Training Plus Mental Training; Train the Brain Model
  Arms: MOTIFS

SUMMARY:
Anterior cruciate ligament injury is a common issue in sports involving cutting and jumping. Treatment may include surgical intervention followed by physical therapy, or no surgical intervention with the main treatment being physical therapy. Despite meeting physical therapist requirements for return to sport, many athletes do not return to sport. This discrepancy in the physical requirements for returning to physical activity and actually returning to the same physical activity level leads to the question of whether current rehabilitation treatments may be improved upon.

One potential method is by integrating mental training into physical rehabilitation. By using mental training and increasing the meaning and relevance of rehabilitation, a person may be preparing more effectively for return to the pace and intensity common during physical activity.

In this study, the investigators aim to create and evaluate a model of training which incorporates physical activity-related movement and mental training in order to more effectively prepare people for return to physical activity after anterior cruciate ligament injury. This will be measured by examining functional hop measures, as well as patient-reported outcomes.

DETAILED DESCRIPTION:
Anterior Cruciate Ligament (ACL) injury is increasingly common in sports involving jumping and cutting. Treatment for such injuries most often includes physical therapist-supervised rehabilitation, with or without surgical reconstruction. Care-as-usual rehabilitation often includes neuromuscular training in order to improve function and reduce knee-related symptoms. Recent data shows that 90% of athletes undergoing rehabilitation achieved normal or nearly-normal knee function when measured in strength and knee laxity. Despite this number, 56% of these athletes did not return to sport or pre-injury activity levels. Due to this imbalance, the question is raised of whether there is a potential to supplement care-as-usual in order to improve upon current rehabilitative training programs.

One attractive alternative is the use of dynamic motor imagery (DMI), which is a form of mental training intended to increase functional equivalence. This is done by imaging an activity-specific and relevant movement while simultaneously completing a similar movement, thereby simulating a real-life physical activity movement. This approach makes it possible to create a situation in which a person is able to create meaning and find relevance in movement used in a rehabilitative training environment.

In this study, the investigators aim to create and test a new training model, referred to as MOTor Imagery to Facilitate Sensorimotor re-learning (MOTIFS), and compare the efficacy of neuromuscular training plus dynamic motor imagery vs neuromuscular training alone in terms of muscle function and patient-reported outcomes in people with an ACL injury and with a goal of returning to pre-injury level of activity.

Primary Hypothesis: 12 weeks of neuromuscular training plus dynamic motor imagery will improve muscle function, measured by relative change in hop performance in the injured leg in side hop test, and patient-reported measures of psychological readiness to return to sport to a greater extent and with a quicker onset of recovery than neuromuscular training alone.

Methods:

In this randomized controlled trial, the inclusion criteria are as follows: (i) male and female ACL-injured people, (ii) over the age of 16, (iii) ACL injury or reconstruction with or without associated injuries to other knee structures, (iii) currently undergoing rehabilitation, (iv) active in recreational or competitive physical activity prior to the injury, and (v) have a goal of reaching pre-injury activity level. Exclusion criteria for participants include: (i) a disease or disorder overriding the knee injury, (ii) have undergone return-to-activity evaluation by a physical therapist, and (iii) do not understand a Scandinavian language (Swedish, Danish, Norwegian) or English.

Those participants randomized to the care-as-usual group will receive rehabilitation according to standard practices.

The experimental group will receive standard training which has been supplemented with the dynamic motor imagery in the MOTIFS model. In this experimental condition, physical therapists will be educated in the use of the new training model and will administer it during clinical practice with the participants. The new model includes information intended to open a dialogue with the participant in order to create a mental simulation in which the participant is able to mentally create a realistic and relevant situation in order to maximize the meaning and motivation of the rehabilitation exercises. This may include the use of sporting equipment, such as balls or sticks, in order to make the rehabilitation session seem as similar to a training session in the relevant sport as possible.

Outcomes:

At baseline and 12 weeks, participants will be measured in patient-reported outcomes, hop ability, and will be filmed in a series of functional tests in order to evaluate postural orientation errors. The main outcomes are relative change in hop performance on the injured leg in a side hop test, and psychological readiness to return to sport (ACL Return to Sport After Injury Scale). Secondary outcomes include a hop test battery (single-leg hop for distance and sidehop), postural orientation errors (single-leg squat, stair descending, forward lunge, side hop, and single-leg hop for distance), Knee Osteoarthritis Outcome Score, Rehabilitation Outcome Satisfaction, Motivation, Patient Enablement Instrument, Physical Activity Enjoyment Scale, and the Tegner Activity scale. A subgroup of both physical therapists and patients will also be asked a series of open-ended questions in a phenomenological interview upon completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Over the age of 16
* Traumatic knee injury with or without surgical intervention, and involving one or more knee structures
* Currently undergoing physical therapist-supervised rehabilitation and have reached the stage in rehabilitation which includes single-leg hop training (i.e. able to complete a side hop and a single-leg hop for distance)
* Active before the injury in recreational or competitive physical activity, with a goal of returning to physical activity

Exclusion Criteria:

* Any degenerative knee disorder, or other disease or disorder overriding the knee injury (e.g. spine disorder, neurological disease)
* Have reached end-stage rehabilitation (i.e. have undergone return to activity evaluation by their physical therapist) or is estimated to return less than 12 weeks from inclusion date
* Do not understand the languages of interest (Swedish, Danish, Norwegian), or English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2018-03-25 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Side Hop | 12 weeks
  Change in hop performance on the injured leg from baseline to 12 weeks, expressed in number of hops completed
Anterior Cruciate Ligament Return to Sport After Injury Scale | 12 months
  12 question self-reported outcome scale measuring readiness to return to sport. Scale ranges from 0-10 for each question. Scores summed from 0 (worst) - 100 (best).

SECONDARY OUTCOMES:
Test Battery to Assess Postural Orientation During Functional Tasks | 12 weeks
  Single-leg Squat, Stair Descending, Forward Lunge, Single-leg hop for distance will be used to evaluate postural orientation by visual film review in which knee medial to foot position is assessed and given a score of either 0 ("good postural orientation" i.e. presents no signs of postural orientation errors), 1 ("fair" i.e. presents signs of postural orientation errors), 2 ("poor" i.e. presents clear signs of postural orientation errors), or 3 ("very poor" i.e. the execution of the test does not have any similarities to the task).
Hop Test Battery | 12 weeks
  Results of side hop and single-leg hop for distance tasks, expressed in percent Limb Symmetry Index (LSI)
Knee Injury and Osteoarthritis Outcome Score | 12 weeks; 12 month follow-up
  Self-reported outcome scale measuring 5 aspects of knee function and symptoms. Subscales include: "Symptoms" - 7 questions; "Pain" - 9 questions; "Function, daily living" - 17 questions; "Function, sports and recreational activities" - 5 questions; "Quality of life" - 4 questions. Responses are given on a 5-point likert scale. Each subscale is given a 0 (extreme symptoms) - 100 (no symptoms) normalized score. A total score will not be presented.
Rehabilitation Outcome Satisfaction | 12 months; 12 month follow-up
  1 self-reported outcome question regarding the satisfaction with rehabilitation. Scores range from 3 ("happy") to -3 ("unhappy").
Perceived Stress Scale | 12 weeks; 12 month follow-up
  Self-reported outcome scale measuring perceived stress. Ten questions on a 5-point likert scale will provide a score from 0 - 40. Score of 0-13 are considered low stress, 14-26 are considered moderate stress, and 27-40 are considered high stress.
Motivation | 12 weeks; 12 month follow-up
  3 questions regarding motivation in regards to return to sport. Scores on a 1 (worst) - 10 (best) scale for each question will be presented individually.
Physical Activity Enjoyment Scale | 12 weeks; 12 month follow-up
  Self-reported outcome scale measuring the perceived enjoyment in an activity. 18 bipolar statements are evaluated on a 7-point likert scale. 11 items are reverse scored. Higher scores indicate greater enjoyment.
Patient Enablement Instrument | 12 weeks
  Self-reported outcome scale measuring the degree of enablement a patient feels (control, understanding, etc) on a 3-point scale where 0 is "not relevant" or "same or less", 1 is "better" and 3 is "much better." The total score is presented as 0-12, with higher scores reflecting higher enablement.
Compliance to intervention in minutes | 12 weeks
  Attendance and participation in rehabilitation activities. Attendance will be reported by the physical therapist (yes/no, minutes). The patient will answer weekly self-reported questions regarding the amount of time engaged in either care as usual or MOTIFS training, both at home and supervised), presented in number of occasions and minutes.
Tegner Activity Scale | 12 months
  Pre-injury, present and final activity level to determine return to sport
Phenomenological Interview | 12 weeks
  Interview regarding subjective experiences of rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
A Study Protocol was published in Trials (DOI: 10.1186/s13063-021-05713-8) October 2021.
  Upon completion of data collection and analysis, data may be available from the author upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Upon completion of data collection (estimated completion January 2022). Data availability in accordance with data management guidelines at Lund University (e.g. available up to 15 years after publication/finalized project)
Access Criteria: Data may be shared upon reasonable request by contacting the corresponding author:
  Niklas Cederström niklas.cederstrom@med.lu.se
URL: https://lucris.lub.lu.se/admin/files/138815992/MOTIFS_Data_Management_Protocol_1.6_2023_02_24.pdf

REFERENCES:
- [Background] Ageberg E, Thomee R, Neeter C, Silbernagel KG, Roos EM. Muscle strength and functional performance in patients with anterior cruciate ligament injury treated with training and surgical reconstruction or training only: a two to five-year followup. Arthritis Rheum. 2008 Dec 15;59(12):1773-9. doi: 10.1002/art.24066. PMID 19035430
- [Background] Frobell RB, Roos EM, Roos HP, Ranstam J, Lohmander LS. A randomized trial of treatment for acute anterior cruciate ligament tears. N Engl J Med. 2010 Jul 22;363(4):331-42. doi: 10.1056/NEJMoa0907797. PMID 20660401
- [Background] Ardern CL, Taylor NF, Feller JA, Webster KE. Fifty-five per cent return to competitive sport following anterior cruciate ligament reconstruction surgery: an updated systematic review and meta-analysis including aspects of physical functioning and contextual factors. Br J Sports Med. 2014 Nov;48(21):1543-52. doi: 10.1136/bjsports-2013-093398. Epub 2014 Aug 25. PMID 25157180
- [Background] Ardern CL, Webster KE, Taylor NF, Feller JA. Return to sport following anterior cruciate ligament reconstruction surgery: a systematic review and meta-analysis of the state of play. Br J Sports Med. 2011 Jun;45(7):596-606. doi: 10.1136/bjsm.2010.076364. Epub 2011 Mar 11. PMID 21398310
- [Background] Risberg MA, Grindem H, Oiestad BE. We Need to Implement Current Evidence in Early Rehabilitation Programs to Improve Long-Term Outcome After Anterior Cruciate Ligament Injury. J Orthop Sports Phys Ther. 2016 Sep;46(9):710-3. doi: 10.2519/jospt.2016.0608. PMID 27581178
- [Background] Guillot A, Moschberger K, Collet C. Coupling movement with imagery as a new perspective for motor imagery practice. Behav Brain Funct. 2013 Feb 20;9:8. doi: 10.1186/1744-9081-9-8. PMID 23425312
- [Background] Smith D, et al. It's All in the Mind: PETTLEP-Based Imagery and Sports Performance. J Appl Sport Psychol 2007;19:80-92.
- [Background] Cumming J, et al. Introducing the revised applied model of deliberate imagery use for sport, dance, exercise, and rehabilitation. Movement & Sport Sciences 2013;1:69-81.
- [Background] Grooms DR, Page SJ, Onate JA. Brain Activation for Knee Movement Measured Days Before Second Anterior Cruciate Ligament Injury: Neuroimaging in Musculoskeletal Medicine. J Athl Train. 2015 Oct;50(10):1005-10. doi: 10.4085/1062-6050-50.10.02. Epub 2015 Sep 29. PMID 26509775
- [Background] Holmes PS, Collins DJ. The PETTLEP approach to motor imagery: A functional equivalence model for sport psychologists. Journal of Applied Sport Psychology 2001;13(1):60-83. doi: 10.1080/104132001753155958
- [Background] Webster KE, Feller JA, Lambros C. Development and preliminary validation of a scale to measure the psychological impact of returning to sport following anterior cruciate ligament reconstruction surgery. Phys Ther Sport. 2008 Feb;9(1):9-15. doi: 10.1016/j.ptsp.2007.09.003. Epub 2007 Nov 5. PMID 19083699
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Background] Gustavsson A, Neeter C, Thomee P, Silbernagel KG, Augustsson J, Thomee R, Karlsson J. A test battery for evaluating hop performance in patients with an ACL injury and patients who have undergone ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2006 Aug;14(8):778-88. doi: 10.1007/s00167-006-0045-6. Epub 2006 Mar 9. PMID 16525796
- [Background] Nae J, Creaby MW, Cronstrom A, Ageberg E. Measurement properties of visual rating of postural orientation errors of the lower extremity - A systematic review and meta-analysis. Phys Ther Sport. 2017 Sep;27:52-64. doi: 10.1016/j.ptsp.2017.04.003. Epub 2017 Apr 18. PMID 28647205
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Howie JG, Heaney DJ, Maxwell M, Walker JJ. A comparison of a Patient Enablement Instrument (PEI) against two established satisfaction scales as an outcome measure of primary care consultations. Fam Pract. 1998 Apr;15(2):165-71. doi: 10.1093/fampra/15.2.165. PMID 9613486
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kendzierski D, DeCarlo KJ. Physical Activity Enjoyment Scale: Two Validation Studies. Journal of Sport and Exercise Psychology 1991;13(1):50-64. doi: 10.1123/jsep.13.1.50
- [Background] Ardern CL, Osterberg A, Sonesson S, Gauffin H, Webster KE, Kvist J. Satisfaction With Knee Function After Primary Anterior Cruciate Ligament Reconstruction Is Associated With Self-Efficacy, Quality of Life, and Returning to the Preinjury Physical Activity. Arthroscopy. 2016 Aug;32(8):1631-1638.e3. doi: 10.1016/j.arthro.2016.01.035. Epub 2016 Mar 24. PMID 27020461
- [Background] Cederstrom N, Graner S, Nilsson G, Ageberg E. Effect of motor imagery on enjoyment in knee-injury prevention and rehabilitation training: A randomized crossover study. J Sci Med Sport. 2021 Mar;24(3):258-263. doi: 10.1016/j.jsams.2020.09.004. Epub 2020 Sep 10. PMID 32958377
- [Background] Cederstrom N, Graner S, Nilsson G, Dahan R, Ageberg E. Motor Imagery to Facilitate Sensorimotor Re-Learning (MOTIFS) after traumatic knee injury: study protocol for an adaptive randomized controlled trial. Trials. 2021 Oct 21;22(1):729. doi: 10.1186/s13063-021-05713-8. PMID 34674738
- [Derived] Cederstrom N, Nilsson G, Dahan R, Graner S, Ageberg E. Using an integrated motor imagery and physical training intervention after knee injury: an interim analysis of the MOTIFS randomised controlled trial. BMJ Open Sport Exerc Med. 2024 Oct 2;10(4):e002064. doi: 10.1136/bmjsem-2024-002064. eCollection 2024. PMID 39371411
- [Derived] Cederstrom N, Ageberg E, Graner S. Lived experiences of patients undergoing treatment for traumatic knee injury using integrated psychological training (MOTIFS) in the context of care-as-usual training: a phenomenological interview study. BMJ Open Sport Exerc Med. 2022 Nov 22;8(4):e001409. doi: 10.1136/bmjsem-2022-001409. eCollection 2022. PMID 36439865
- Available data/document: Statistical Analysis Plan — https://lucris.lub.lu.se/admin/files/138815992/MOTIFS_Data_Management_Protocol_1.6_2023_02_24.pdf